CLINICAL TRIAL: NCT06202625
Title: Efficacy and Safety of Avatrombopag in the Treatment of Thrombocytopenia After Haploidentical Hematopoietic Stem Cell Transplantation: Prospective, Multi-center, Double-blinded, Randomized Placebo-controlled Study
Brief Title: Efficacy and Safety of Avatrombopag in the Treatment of Thrombocytopenia After Haplo-HSCT
Acronym: Haplo-HSCT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Xiangya Hospital of Central South University (Other); Sichuan Provincial People's Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Shanxi Bethune Hospital (Other); 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other); Tang-Du Hospital (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023PHD009-001
Record Dates: First submitted 2023-12-14; First posted 2024-01-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Thrombocytopenia; Stem Cell Transplant Complications
Keywords: Thrombocytopenia; hematopoietic stem cell transplantation; haploidentical
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- avatrombopag (Experimental): Avatrombopag 20 mg/d will be taken orally from +D7 after haplo-HSCT until reaching the adjustment indication or to +D60 after haplo-HSCT. Routine treatment is allowed.
  Adjustment indication:
  When PLT<50×10^9/L or PLT transfusion dependent on the +D30 after haplo-HSCT, increase the dosage to 40 mg/d; When the dosage has been increased to 40 mg/d, and PLT≥80×10^9/L excluding the factor of PLT transfusion, decrease the dosage to 20 mg/d; When PLT≥80×10^9/L for 7 consecutive days excluding the factor of PLT transfusion, or PLT≥300×10^9/L excluding the factor of PLT transfusion, stop administration; When PLT<50×10^9/L or become PLT transfusion dependent after stopping administration, initiate administration again at the dosage 40 mg/d.
  PLT transfusion Indication: When PLT<20×10^9/L, and/or with the symptom or risk of bleeding.
  Interventions: Drug: avatrombopag
- Placebo (Placebo Comparator): Placebo 20 mg/d will be taken orally from +D7 after haplo-HSCT until reaching the adjustment indication or to +D60 after haplo-HSCT. Routine treatment is allowed.
  Adjustment indication:
  When PLT<50×10^9/L or PLT transfusion dependent on the +D30 after haplo-HSCT, increase the dosage to 40 mg/d; When the dosage has been increased to 40 mg/d, and PLT≥80×10^9/L excluding the factor of PLT transfusion, decrease the dosage to 20 mg/d; When PLT≥80×10^9/L for 7 consecutive days excluding the factor of PLT transfusion, or PLT≥300×10^9/L excluding the factor of PLT transfusion, stop administration; When PLT<50×10^9/L or become PLT transfusion dependent after stopping administration, initiate administration again at the dosage 40 mg/d.
  PLT transfusion Indication: When PLT<20×10^9/L, and/or with the symptom or risk of bleeding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: avatrombopag — The avatrombopag 20mg/d will be orally taken from +D7 after haplo-HSCT until meeting the adjustment indication or to +D60 after haplo-HSCT; When PLT<50×10^9/L or PLT transfusion-dependent on the +D30 after haplo-HSCT, increase avatrombopag dosage to 40 mg/d; When PLT≥80×10^9/L and without PLT transfusion within avatrombopag dosage at 40 mg/d, decrease avatrombopag dosage to 20 mg/d; When PLT≥80×10^9/L for 7 consecutive days or PLT≥300×10^9/L and without PLT transfusion, stop avatrombopag; When PLT<50×10^9/L or PLT transfusion-dependent after stopping avatrombopag , reuse avatrombopag at 40 mg/d.
  Other Names: Doptelet
  Arms: avatrombopag
Drug: Placebo — The placebo 20mg/d will be orally taken from +D7 after haplo-HSCT until meeting the adjustment indication or to +D60 after haplo-HSCT; When PLT<50×10^9/L or PLT transfusion-dependent on the +D30 after haplo-HSCT, increase placebo dosage to 40 mg/d; When PLT≥80×10^9/L and without PLT transfusion within placebo dosage at 40 mg/d, decrease placebo dosage to 20 mg/d; When PLT≥80×10^9/L for 7 consecutive days or PLT≥300×10^9/L and without PLT transfusion, stop placebo; When PLT<50×10^9/L or PLT transfusion-dependent after stopping placebo, reuse placebo at 40 mg/d.
  Arms: Placebo

SUMMARY:
In this study, investigators aim to evaluate the efficacy of avatrombopag in thrombocytopenic patients after haploidentical hematopoietic stem cell transplantation (haplo-HSCT) through a prospective, multi-center, double-blinded, randomized placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Thrombocytopenia is a common and severe complication after haplo-HSCT, including primary isolated thrombocytopenia (PIT) and secondary failure of platelet recovery (SFPR), which may cause bleeding and infection, and thus influence the OS, DFS, and NRM of the patients. Avatrombopag has been proved effective and safe in patients with chronic liver disease(CLD) and immune thrombocytopenia (ITP) and have been approved for CLD-associated thrombocytopenia undergoing elective invasive procedure (FDA&NMPA) and ITP(FDA). Chinese consensus has recommended avatrombopag and some other thrombopoietin receptor agonists (TPO-RAs) to treat thrombocytopenia after haplo-HSCT. However, it lacks prospective studies to support that.Investigators aim to evaluate the efficacy of avatrombopag in thrombocytopenic patients after haplo-HSCT through a prospective, multi-center, double-blinded, randomized placebo-controlled clinical trial.

The patients with PLT<20×10^9/L or transfusion dependent on the 7th day (+D7) after haplo-HSCT are included and assigned in a 1:1 randomization schedule to the avatrombopag group (receiving avatrombopag, n=71）and the placebo group (receiving placebo, n=71). The primary endpoint is the proportion of participants whose PLT≥50×10^9/L on +D60 after haplo-HSCT without the need for PLT transfusion for 7 consecutive days or above. Second endpoints includ the proportion of participants whose PLT≥100×10^9/L on +D60 after haplo-HSCT without the need for PLT transfusion for 7 consecutive days or above, the proportion of participants whose PLT≥20×10^9/L and whose PLT≥50×10^9/L on +D30 after haplo-HSCT without the need for PLT transfusion for 7 consecutive days or above, the proportion of participants whose PLT≥50×10^9/L and whose PLT≥100×10^9/L on +D90 after haplo-HSCT without the need for PLT transfusion for 7 consecutive days or above, the first day to achieve PLT≥20×10^9/L and PLT≥50×10^9/L and PLT≥100×10^9/L without the need for PLT transfusion for consecutive 7 days and above within +D60 after haplo-HSCT, the percentage of participants who need PLT transfusion and the average count of PLT from +D7 to + D60 after haplo-HSCT, the first day and the percentage of participants to achieve absolute neutrophil≥500/μL for consecutive 3 days within +D30 after haplo-HSCT, the graft-versus-host disease(GVHD), infection, the overall survival(OS),the disease free survival(DFS) and the non-relapse mortality(NRM) rates of participants within the first year after haplo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18-65 years;
2. PLT<20×10^9/L or transfusion dependent on +D7 after haplo-HSCT;
3. Agree to receive the treatment of avatrombopag after Haplo-HSCT and sign the informed consent form.

Exclusion Criteria:

1. With active infection;
2. ALT or AST>3ULN, or total Bil>2ULN
3. Ccr<50 mL/min;
4. With the history of arteriovenous thrombosis;
5. With history of cardiovascular disease (such as NYHA Class III/IV congestive heart failure, arrhythmia that increases the risk of thromboembolic events [such as atrial fibrillation] and angina), and subjects who have undergone coronary stent implantation, angioplasty, or coronary artery bypass grafting;
6. With treatment of drugs to promote platelet production two weekes before enrollment, including but not limited to rhTPO and TPO-RA;
7. HBsAg or anti-HCV or anti-HIV positive;
8. Known to be allergic to avatrombopag and any of its excipients;
9. With secondary or multiple HSCT;
10. Females who were pregnant or breastfeeding or who had fertile ability but refuse to take effective contraceptive measures during and one month after this trial;
11. With any other clinical trial of investigational product or device within 30 days prior to the baseline visit, except for observational study;
12. Deemed unsuitable for enrollment by the investigator for any history of or concomitant medical condition.
13. Concomitant medication:The rhIL-11, rhTPO or TPO-RA(such as eltrombopag, hetrombopag and romiplostim) and desitabine, etc. were not allowed for use during this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of complete response(CR) on day 60 after haplo-HSCT | from randomization to day 60 after haplo-HSCT
  the proportion of participants whose PLT≥50×10^9/L on day 60 after haplo-HSCT independent of PLT transfusion for 7 consecutive days or above

SECONDARY OUTCOMES:
the proportion of resonse(R)/remission on day 60 after haplo-HSCT | from randomization to day 60 after haplo-HSCT
  the proportion of participants whose PLT≥20×10^9/L or PLT≥100×10^9/L on day 60 after haplo-HSCT independent of PLT transfusion for 7 consecutive days or above
the proportion of R/CR on day 30 after haplo-HSCT | from randomization to day 30 after haplo-HSCT
  the proportion of participants whose PLT≥20×10^9/L or PLT≥50×10^9/L on day 30 after haplo-HSCT independent of PLT transfusion for 7 consecutive days or above,respectively
the proportion of CR/remission on day 90 after haplo-HSCT | from randomization to day 90 after haplo-HSCT
  the proportion of participants whose PLT≥50×10^9/L or PLT≥100×10^9/L on day 90 after haplo-HSCT independent of PLT transfusion for 7 consecutive days or above
Time to R/CR/remission | from randomization to day 60 after haplo-HSCT
  the first day of the time to achieve PLT≥20×10^9/L and PLT≥50×10^9/L or PLT≥100×10^9/L independent of PLT transfusion for consecutive 7 days and above within 60 days after haplo-HSCT,respectively
PLT transfusion dependence | from randomization to day 60 after haplo-HSCT
  the percentage of participants who need PLT transfusion and the average volume of transfused PLT from day 7 to day 60 after haplo-HSCT
neutrophil engraftment | from randomization to day 30 after haplo-HSCT
  the first day and the percentage of participants to achieve absolute neutrophil≥500/μL for consecutive 3 days within 30 days after haplo-HSCT
GVHD | from randomization to 1 year after haplo-HSCT
  the incidece of graft versus host disease(GVHD)
overall survival(OS) | from randomization to 1 year after haplo-HSCT
  the 1-year OS of participants
disease free survival(DFS) | from randomization to 1 year after haplo-HSCT
  the 1-year DFS of participants
non-relapse mortality(NRM) | from randomization to 1 year after haplo-HSCT
  the 1-year NRM of participants

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, Principal Investigator — Peking University People's Hospital
Locations (14):
- China (14):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Guangzhou First People's Hospital, School of Medicine, South China University of Technology, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital, Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanxi Tumor Hospital Affiliated to Shanxi Medical University, Taiyuan, Shanxi
  - Tangdu Hospital, PLA Air Force Military Medical University, Xi’an, Shanxi
  - Xinqiao Hospital, Army Military Medical University, Chongqing, Sichuan
  - 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan
  - Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin